CLINICAL TRIAL: NCT01640951
Title: A Multicenter, Double-blind and Open Label, 4 Year Extension Study of Subcutaneous Secukinumab in Prefilled Syringes, Assessing Long-term Safety, Tolerability and Efficacy in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis Treated With Either a Fixed Dose Regimen or on a Retreatment at Start of Relapse Regimen
Brief Title: 4 Year Extension Study of Efficacy and Safety of Secukinumab in Patients With Moderate to Severe Chronic Plaque-type Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2304E1; 2012-000985-39 (EudraCT Number)
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-04

CONDITIONS: Moderate to Severe Chronic Plaque-Type Psoriasis
Keywords: Psoriasis; Plaque; Inflammatory skin disease; Scaly patches; AIN457; Secukinumab; Moderate to Severe Plaque-type Psoriasis
MeSH Terms: conditions — Psoriasis; Plaque, Amyloid; Dermatitis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- AIN457 150 mg - Fixed Interval (FI) (Experimental): 1 s.c. Secukinumab 150 mg Pre-filled seringue (PFS) injection + 1 s.c. Placebo (PBO) Secukinumab PFS injection every 4 weeks
  Interventions: Drug: AIN457 150 mg; Drug: Placebo
- AIN457 150 mg - Start of relapse (SoR) (Experimental): Start of relapse: 1 s.c. Secukinumab 150 mg PFS injection + 1 s.c. PBO Secukinumab PFS injection every 4 weeks
  Otherwise: 2 s.c. PBO Secukinumab PFS injections every 4 weeks
  Interventions: Drug: AIN457 150 mg; Drug: Placebo
- AIN457 300 mg - Fixed Interval (FI) (Experimental): 2 s.c. Secukinumab 150 mg PFS injections every 4 weeks
  Interventions: Drug: AIN457 300 mg
- AIN457 300 mg - Start of Relapse (SoR) (Experimental): Start of relapse: 2 s.c. Secukinumab 150 mg PFS injection every 4 weeks
  Otherwise: 2 s.c. PBO Secukinumab PFS injections every 4 weeks
  Interventions: Drug: AIN457 300 mg; Drug: Placebo
- AIN457 300 mg - Open Label (OL) (Experimental): Open Label - Secukinumab 300mg every 4 weeks
  Interventions: Drug: AIN457 300 mg

INTERVENTIONS:
Drug: AIN457 150 mg — (1 injection per dose) and placebo to Secukinumab 150 mg
  Other Names: Secukinumab 150 mg
  Arms: AIN457 150 mg - Fixed Interval (FI); AIN457 150 mg - Start of relapse (SoR)
Drug: AIN457 300 mg — Secukinumab 150 mg (2 injections per dose)
  Other Names: Secukinumab 300 mg
  Arms: AIN457 300 mg - Fixed Interval (FI); AIN457 300 mg - Open Label (OL); AIN457 300 mg - Start of Relapse (SoR)
Drug: Placebo
  Arms: AIN457 150 mg - Fixed Interval (FI); AIN457 150 mg - Start of relapse (SoR); AIN457 300 mg - Start of Relapse (SoR)

SUMMARY:
CAIN457A2304E1 was an extension study to two phase III studies, CAIN457A2304 and CAIN457A2307 (core studies). This extension study planned to collect up to four years of long-term safety, tolerability and efficacy data of secukinumab in both the fixed interval regimen and the retreatment at start of relapse regimen. All subjects who completed the full study treatment period (52 weeks) in the cores studies CAIN457A2304 and CAIN457A2307 were eligible to participate in this extension study. In this extension study, the prefilled syringe (PFS) liquid formulation of secukinumab was used.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to understand and communicate with the investigator and comply with the requirements of the study and must give a written, signed and dated informed consent before any study related activity is performed. Where relevant, a legal representative will also sign the informed consent according to local laws and regulations.
2. Subjects who complete Week 52 of study CAIN457A2304 or complete Week 40 of study CAIN457A2307
3. Subjects expected to benefit from participation in the extension study, as assessed by the subject and investigator

Exclusion Criteria:

1. A protocol deviation in the core studies which according to the investigator will prevent the meaningful analysis of the extension study for the individual subject
2. Ongoing use of prohibited psoriasis or non-psoriasis treatments. Time period from last use of prohibited treatments in the core study to first dose of study drug in this extension study.
3. Subjects expected to be exposed to an undue safety risk if participating in the trial
4. Current severe progressive or uncontrolled disease which in the judgment of the investigator renders the subject unsuitable for the trial
5. Plans for administration of live vaccines during the study period
6. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>10 mIU/mL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2012-09-16 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (102):
- United States (27):
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Champaign, Illinois
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Fridley, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Verona, New Jersey
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Anderson, South Carolina
  - Novartis Investigative Site, Greer, South Carolina
  - Novartis Investigative Site, Goodlettsville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
- Novartis Investigative Site, Wels, Austria
- Bulgaria (3):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (5):
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, Oakville, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Czechia (6):
  - Novartis Investigative Site, Brno-Bohunice, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Prague, CZE
  - Novartis Investigative Site, České Budějovice
  - Novartis Investigative Site, Nový Jičín
  - Novartis Investigative Site, Prague
- France (5):
  - Novartis Investigative Site, Antony
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Toulouse
- Germany (18):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Bad Wildbad
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Buchholz I. D. Nordheide
  - Novartis Investigative Site, Dippoldiswalde-Schmiedeberg
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mahlow
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Wuppertal
- Italy (3):
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Verona, VR
- Japan (14):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kisarazu, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Poland (3):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (5):
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Svidník
  - Novartis Investigative Site, Žilina
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- United Kingdom (5):
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Blackpool
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Poole
- Vietnam (3):
  - Novartis Investigative Site, Ho Chi Minh City, VNM
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Bissonnette R, Luger T, Thaci D, Toth D, Messina I, You R, Guana A, Fox T, Papavassilis C, Gilloteau I, Mrowietz U. Secukinumab sustains good efficacy and favourable safety in moderate-to-severe psoriasis after up to 3 years of treatment: results from a double-blind extension study. Br J Dermatol. 2017 Oct;177(4):1033-1042. doi: 10.1111/bjd.15706. Epub 2017 Sep 4. PMID 28580579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 675 subjects from the core studies (CAIN457A2304 and CAIN457A2307) were enrolled at 112 sites. Subjects enrolled in the secukinumab 300 mg Open-Label (OL) arm came only from the CAIN457A2307 study, as such they were partial responders at Week 12, while all other subjects in the extension were PASI 75 responders at Week 12 in the core study.
Pre-assignment Details: At Week 156, subjects who rolled over from the CAIN457A2304 study were unblinded and provided an option to switch to one of the treatment options described below upon investigator judgment; subjects from the CAIN457A2307 study could administer study drug at home every 4 weeks, but were required to come for office visits every 12-16 weeks.
Groups:
- AIN150FI: AIN457 150 mg - Fixed Interval (FI)
- AIN150 FI_AIN300 FI: AIN457 150 mg FI switch to AIN457 300 mg FI (150 mg FI SW)
- AIN300 FI: AIN457 300 mg - Fixed Interval (FI)
- AIN150 SoR: AIN457 150 mg - Start of Relapse (SoR)
- AIN150 SOR_AIN300 FI: AIN457 150 mg SoR switch to AIN457 300 mg FI (150 mg SoR SW)
- AIN300 SoR: AIN457 300 mg - Start of Relapse (SoR)
- AIN300 SoR _ AIN300 FI: AIN457 300 mg SoR switch to AIN457 300 mg FI (300 mg SoR SW)
- AIN300 OL: AIN457 300 mg Open-label (OL)
Period: Overall Study
Arm/Group | AIN150FI | AIN150 FI_AIN300 FI | AIN300 FI | AIN150 SoR | AIN150 SOR_AIN300 FI | AIN300 SoR | AIN300 SoR _ AIN300 FI | AIN300 OL
Started (All randomized patients (Full Analysis Set and Safety Set)) | 77 | 75 | 168 | 55 | 95 | 60 | 112 | 33
Completed | 31 | 60 | 126 | 10 | 82 | 13 | 94 | 17
Not Completed | 46 | 15 | 42 | 45 | 13 | 47 | 18 | 16
Not completed — Adverse Event | 8 | 3 | 10 | 6 | 1 | 11 | 1 | 3
Not completed — Lack of Efficacy | 20 | 1 | 7 | 14 | 0 | 6 | 5 | 6
Not completed — Lost to Follow-up | 1 | 0 | 6 | 2 | 2 | 3 | 1 | 1
Not completed — Non-compliance with study treatment | 0 | 0 | 1 | 1 | 1 | 4 | 1 | 0
Not completed — Physician Decision | 2 | 5 | 2 | 2 | 2 | 3 | 3 | 0
Not completed — Pregnancy | 3 | 0 | 0 | 4 | 0 | 0 | 2 | 0
Not completed — Protocol Deviation | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Not completed — Subject/Guardian decision | 12 | 4 | 13 | 15 | 7 | 19 | 5 | 4
Not completed — Death | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN150FI | AIN150 FI_AIN300 FI | AIN300 FI | AIN150 SoR | AIN150 SOR_AIN300 FI | AIN300 SoR | AIN300 SoR _ AIN300 FI | AIN300 OL | Total
Number analyzed (Participants) | 77 | 75 | 168 | 55 | 95 | 60 | 112 | 33 | 675
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (13.24) | 46.0 (12.03) | 48.5 (12.54) | 42.7 (12.23) | 48.0 (12.13) | 45.2 (12.08) | 44.6 (13.09) | 46.5 (13.99) | 45.9 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 25 | 50 | 25 | 28 | 18 | 35 | 12 | 231
  Male | 39 | 50 | 118 | 30 | 67 | 42 | 77 | 21 | 444
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 13 | 14 | 31 | 5 | 21 | 9 | 26 | 4 | 123
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 2 | 1 | 2 | 0 | 3 | 3 | 1 | 0 | 12
  White | 62 | 60 | 132 | 48 | 68 | 45 | 84 | 29 | 528
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 3 | 2 | 1 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Long-term Safety and Tolerability of Secukinumab
Description: Analysis of absolute and relative frequencies for treatment emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths by primary System Organ Class (SOC)
Time Frame: Week 268
Population: Safety Set. All subjects who took at least one dose of study treatment during the extension treatment period. A subject with multiple adverse events within a primary system organ class was counted only once in the total row. Deaths up to 28 days after the last dose are included. Only descriptive analysis done.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN150FI | AIN150 FI_AIN300 FI | AIN300 FI | AIN150 SoR | AIN150 SOR_AIN300 FI | AIN300 SoR | AIN300 SoR _ AIN300 FI | AIN300 OL
Number analyzed (Participants) | 77 | 75 | 168 | 55 | 95 | 60 | 112 | 33
Percentage of participants
  AEs by Primary System Organ Class (SOC) | 88.3 | 92.0 | 92.9 | 78.2 | 87.4 | 80.0 | 94.6 | 93.9
  SAEs by Primary System Organ Class (SOC) | 20.8 | 24.0 | 23.8 | 16.4 | 20.0 | 18.3 | 17.0 | 36.4
  Deaths by Primary System Organ Class (SOC) | 0.0 | 1.3 | 0.6 | 0.0 | 0.0 | 0.0 | 0.0 | 6.1

2. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) Score of 75 at Weeks 52, 104, 156, 208 and 260
Description: PASI: Combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4)
Time Frame: Week 52, Week 104, Week 156, Week 208, Week 260
Population: The full analysis set (FAS), which consisted of all participants with an observed value, was considered. Only patients with evaluable data at each time point were analyzed for that time point. Only descriptive analysis done.
Measure: Number; unit: Percentage of Participants
Groups:
- AIN150FI (NSW+SW): AIN457 150 mg - Fixed Interval combined non-switch and switch
Arm/Group | AIN150FI | AIN150 FI_AIN300 FI | AIN150FI (NSW+SW) | AIN300 FI | AIN150 SoR | AIN150 SOR_AIN300 FI | AIN300 SoR | AIN300 SoR _ AIN300 FI | AIN300 OL
Number analyzed (Participants) | 77 | 75 | 152 | 168 | 55 | 95 | 60 | 112 | 33
Percentage of Participants
  Week 52: number analyzed (Participants) | 76 | 75 | 151 | 162 | 55 | 95 | 58 | 111 | 33
  Week 52 | 69.7 | 65.3 | 67.5 | 88.9 | 38.2 | 38.9 | 51.7 | 39.6 | 63.6
  Week 104: number analyzed (Participants) | 60 | 73 | 133 | 152 | 30 | 94 | 34 | 110 | 30
  Week 104 | 63.3 | 54.8 | 58.6 | 80.9 | 40.0 | 39.4 | 55.9 | 44.5 | 63.3
  Week 156: number analyzed (Participants) | 40 | 75 | 115 | 139 | 16 | 94 | 20 | 111 | 21
  Week 156 | 85.0 | 49.3 | 61.7 | 78.4 | 62.5 | 35.1 | 65.0 | 41.4 | 57.1
  Week 208: number analyzed (Participants) | 35 | 69 | 104 | 132 | 11 | 87 | 12 | 100 | 21
  Week 208 | 80.0 | 78.3 | 78.8 | 87.9 | 63.6 | 87.4 | 41.7 | 79.0 | 61.9
  Week 260: number analyzed (Participants) | 29 | 56 | 85 | 122 | 10 | 79 | 13 | 87 | 16
  Week 260 | 89.7 | 71.4 | 77.6 | 88.5 | 50.0 | 86.1 | 53.8 | 81.6 | 75.0

3. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) Scores of 50, 90 and 100 Over Time at Weeks 52, 104, 156, 208 and 260
Description: as for outcome 2
Time Frame: Week 52, Week 104, Week 156, Week 208, Week 260
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN150FI | AIN150 FI_AIN300 FI | AIN150FI (NSW+SW) | AIN300 FI | AIN150 SoR | AIN150 SOR_AIN300 FI | AIN300 SoR | AIN300 SoR _ AIN300 FI | AIN300 OL
Number analyzed (Participants) | 77 | 75 | 152 | 168 | 55 | 95 | 60 | 112 | 33
Percentage of Participants
  Week 52 / PASI 50: number analyzed (Participants) | 76 | 75 | 151 | 162 | 55 | 95 | 58 | 111 | 33
  Week 52 / PASI 50 | 89.5 | 98.7 | 94.0 | 98.8 | 80.0 | 86.3 | 91.4 | 88.3 | 93.9
  Week 52 / PASI 90: number analyzed (Participants) | 76 | 75 | 151 | 162 | 55 | 95 | 58 | 111 | 33
  Week 52 / PASI 90 | 61.8 | 38.7 | 50.3 | 68.5 | 12.7 | 11.6 | 19.0 | 12.6 | 39.4
  Week 52 / PASI 100: number analyzed (Participants) | 76 | 75 | 151 | 162 | 55 | 95 | 58 | 111 | 33
  Week 52 / PASI 100 | 31.6 | 16.0 | 23.8 | 43.8 | 3.6 | 2.1 | 8.6 | 3.6 | 9.1
  Week 104 / PASI 50: number analyzed (Participants) | 60 | 73 | 133 | 152 | 30 | 94 | 34 | 110 | 30
  Week 104 / PASI 50 | 88.3 | 84.9 | 86.5 | 96.7 | 80.0 | 87.2 | 88.2 | 85.5 | 86.7
  Week 104 / PASI 90: number analyzed (Participants) | 60 | 73 | 133 | 152 | 30 | 94 | 34 | 110 | 30
  Week 104 / PASI 90 | 46.7 | 23.3 | 33.8 | 64.5 | 16.7 | 9.6 | 14.7 | 18.2 | 26.7
  Week 104 / PASI 100: number analyzed (Participants) | 60 | 73 | 133 | 152 | 30 | 94 | 34 | 110 | 30
  Week 104 / PASI 100 | 28.3 | 6.8 | 16.5 | 43.4 | 10.0 | 1.1 | 5.9 | 4.5 | 13.3
  Week 156 / PASI 50: number analyzed (Participants) | 40 | 75 | 115 | 139 | 16 | 94 | 20 | 111 | 21
  Week 156 / PASI 50 | 100.0 | 86.7 | 91.3 | 97.1 | 93.8 | 88.3 | 85.0 | 90.1 | 90.5
  Week 156 / PASI 90: number analyzed (Participants) | 40 | 75 | 115 | 139 | 16 | 94 | 20 | 111 | 21
  Week 156 / PASI 90 | 60.0 | 17.3 | 32.2 | 61.9 | 31.3 | 10.6 | 30.0 | 10.8 | 28.6
  Week 156 / PASI 100: number analyzed (Participants) | 40 | 75 | 115 | 139 | 16 | 94 | 20 | 111 | 21
  Week 156 / PASI 100 | 45.0 | 8.0 | 20.9 | 41.7 | 6.3 | 4.3 | 0.0 | 3.6 | 19.0
  Week 208 / PASI 50: number analyzed (Participants) | 35 | 69 | 104 | 132 | 11 | 87 | 12 | 100 | 21
  Week 208 / PASI 50 | 100.0 | 97.1 | 98.1 | 97.0 | 72.7 | 98.9 | 100.0 | 95.0 | 95.2
  Week 208 / PASI 90: number analyzed (Participants) | 35 | 69 | 104 | 132 | 11 | 87 | 12 | 100 | 21
  Week 208 / PASI 90 | 51.4 | 49.3 | 50.0 | 65.9 | 27.3 | 64.4 | 16.7 | 53.0 | 23.8
  Week 208 / PASI 100: number analyzed (Participants) | 35 | 69 | 104 | 132 | 11 | 87 | 12 | 100 | 21
  Week 208 / PASI 100 | 28.6 | 20.3 | 23.1 | 43.2 | 9.1 | 23.0 | 0.0 | 24.0 | 23.8
  Week 260 / PASI 50: number analyzed (Participants) | 29 | 56 | 85 | 122 | 10 | 79 | 13 | 87 | 16
  Week 260 / PASI 50 | 100.0 | 96.4 | 97.6 | 97.5 | 100.0 | 97.5 | 100.0 | 93.1 | 87.5
  Week 260 / PASI 90: number analyzed (Participants) | 29 | 56 | 85 | 122 | 10 | 79 | 13 | 87 | 16
  Week 260 / PASI 90 | 51.7 | 46.4 | 48.2 | 66.4 | 30.0 | 57.0 | 7.7 | 54.0 | 43.8
  Week 260 / PASI 100: number analyzed (Participants) | 29 | 56 | 85 | 122 | 10 | 79 | 13 | 87 | 16
  Week 260 / PASI 100 | 31.0 | 17.9 | 22.4 | 41.0 | 10.0 | 29.1 | 7.7 | 18.4 | 25.0

4. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Weeks 52, 104, 156, 208 and 260
Description: as for outcome 2
Time Frame: Baseline, Week 52, Week 104, Week 156, Week 208, Week 260
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | AIN150FI | AIN150 FI_AIN300 FI | AIN150FI (NSW+SW) | AIN300 FI | AIN150 SoR | AIN150 SOR_AIN300 FI | AIN300 SoR | AIN300 SoR _ AIN300 FI | AIN300 OL
Number analyzed (Participants) | 77 | 75 | 152 | 168 | 55 | 95 | 60 | 112 | 33
Percent change
  Week 52: number analyzed (Participants) | 76 | 75 | 151 | 162 | 55 | 95 | 58 | 111 | 33
  Week 52 | -83.54 (21.744) | -81.47 (16.179) | -82.51 (19.147) | -91.14 (13.377) | -65.13 (23.452) | -67.91 (21.521) | -75.63 (16.970) | -69.13 (18.976) | -79.75 (17.045)
  Week 104: number analyzed (Participants) | 60 | 73 | 133 | 152 | 30 | 94 | 34 | 110 | 30
  Week 104 | -78.13 (26.278) | -72.47 (24.099) | -75.02 (25.168) | -88.48 (16.273) | -63.17 (28.596) | -68.40 (18.057) | -67.62 (40.039) | -70.98 (19.720) | -76.10 (19.342)
  Week 156: number analyzed (Participants) | 40 | 75 | 115 | 139 | 16 | 94 | 20 | 111 | 21
  Week 156 | -90.27 (11.543) | -71.48 (19.892) | -78.02 (19.576) | -88.34 (15.555) | -78.97 (16.709) | -68.71 (18.094) | -77.40 (18.714) | -69.77 (18.586) | -76.12 (20.437)
  Week 208: number analyzed (Participants) | 35 | 69 | 104 | 132 | 11 | 87 | 12 | 100 | 21
  Week 208 | -87.60 (12.296) | -85.06 (14.082) | -85.91 (13.501) | -90.46 (14.116) | -72.64 (24.394) | -89.36 (12.978) | -74.38 (13.817) | -85.25 (17.018) | -79.12 (16.827)
  Week 260: number analyzed (Participants) | 29 | 56 | 85 | 122 | 10 | 79 | 13 | 87 | 16
  Week 260 | -88.75 (10.928) | -84.10 (15.012) | -85.68 (13.867) | -90.06 (14.639) | -76.20 (17.418) | -89.40 (12.763) | -78.13 (10.197) | -85.48 (17.116) | -81.47 (21.335)

5. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment Modified 2011 (IGA) 2011 Score of 0 or 1 Over Time at Weeks 52, 104, 156, 208 and 260
Description: The IGA mod 2011 is a static scale, i.e., it refers exclusively to the participant's disease state at the time of the assessments and does not attempt a comparison to any of the participant's previous disease states at prior visits. The score ranges from 0 (clear) to 4 (severe). The score 0 is clear, 1 is almost clear, 2 is mild, 3 is moderate, and 4 is severe.
Time Frame: Week 52, Week 104, Week 156, Week 208, Week 260
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN150FI | AIN150 FI_AIN300 FI | AIN150FI (NSW+SW) | AIN300 FI | AIN150 SoR | AIN150 SOR_AIN300 FI | AIN300 SoR | AIN300 SoR _ AIN300 FI | AIN300 OL
Number analyzed (Participants) | 77 | 75 | 152 | 168 | 55 | 95 | 60 | 112 | 33
Percentage of Participants
  Week 52 / IGA 0/1: number analyzed (Participants) | 76 | 75 | 151 | 165 | 55 | 95 | 60 | 111 | 33
  Week 52 / IGA 0/1 | 59.2 | 50.7 | 55.0 | 69.1 | 20.0 | 20.0 | 28.3 | 19.8 | 42.4
  Week 104 / IGA 0/1: number analyzed (Participants) | 60 | 73 | 133 | 152 | 30 | 94 | 34 | 110 | 30
  Week 104 / IGA 0/1 | 51.7 | 30.1 | 39.8 | 66.4 | 20.0 | 16.0 | 17.6 | 17.3 | 23.3
  Week 156 / IGA 0/1: number analyzed (Participants) | 40 | 75 | 115 | 139 | 16 | 94 | 20 | 111 | 21
  Week 156 / IGA 0/1 | 62.5 | 21.3 | 35.7 | 56.8 | 37.5 | 14.9 | 25.0 | 15.3 | 28.6
  Week 208 / IGA 0/1: number analyzed (Participants) | 35 | 68 | 103 | 132 | 12 | 87 | 12 | 100 | 21
  Week 208 / IGA 0/1 | 57.1 | 47.1 | 50.5 | 62.1 | 41.7 | 63.2 | 8.3 | 52.0 | 23.8
  Week 260 / IGA 0/1: number analyzed (Participants) | 29 | 56 | 85 | 120 | 10 | 79 | 13 | 87 | 16
  Week 260 / IGA 0/1 | 55.2 | 48.2 | 50.6 | 65.0 | 40.0 | 58.2 | 30.8 | 54.0 | 37.5

6. Secondary Outcome: Percentage Change From Baseline in Dermatology Life Quality Index (DLQI©) Response at Weeks 52, 104, 156, 208 and 260
Description: The DLQI is a quality of life measure used in the psoriatic The 10-item questionnaire has a score range of 0 (best) to 30 (worst) with higher scores indicating poor quality of life. The instrument contains six functional scales (i.e., symptoms and feeling, daily activities, leisure, work and school, personal relationships, treatment). Each item has 4 response categories, ranging from 0 (not at all) to 3 (very much). "Not relevant" is also a valid response and is scored as 0. The DLQI total score is a sum of the 10 questions
Time Frame: Baseline, Week 52, Week 104, Week 156, Week 208, Week 260
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | AIN150FI | AIN150 FI_AIN300 FI | AIN150FI (NSW+SW) | AIN300 FI | AIN150 SoR | AIN150 SOR_AIN300 FI | AIN300 SoR | AIN300 SoR _ AIN300 FI | AIN300 OL
Number analyzed (Participants) | 77 | 75 | 152 | 168 | 55 | 95 | 60 | 112 | 33
Percent change
  Week 52: number analyzed (Participants) | 77 | 74 | 151 | 164 | 54 | 95 | 60 | 108 | 33
  Week 52 | -77.3 [-87.5 to -68.3] | -85.7 [-90.0 to -77.8] | -81.8 [-87.5 to -75.0] | -93.3 [-95.5 to -90.3] | -65.0 [-74.7 to -55.6] | -68.2 [-75.0 to -61.0] | -66.7 [-75.0 to -52.9] | -72.8 [-79.0 to -65.0] | -79.2 [-89.6 to -65.0]
  Week 104: number analyzed (Participants) | 66 | 71 | 137 | 152 | 33 | 91 | 40 | 103 | 29
  Week 104 | -70.8 [-83.3 to -63.3] | -73.8 [-80.4 to -65.9] | -73.3 [-78.1 to -67.3] | -87.5 [-93.3 to -83.3] | -71.9 [-80.2 to -58.6] | -63.6 [-70.8 to -56.3] | -68.8 [-78.9 to -51.8] | -74.9 [-81.2 to -66.7] | -77.2 [-88.9 to -62.0]
  Week 156: number analyzed (Participants) | 39 | 74 | 113 | 137 | 15 | 93 | 21 | 107 | 22
  Week 156 | -89.3 [-97.4 to -81.0] | -67.9 [-75.0 to -60.0] | -75.0 [-80.0 to -69.3] | -91.7 [-93.8 to -86.4] | -79.6 [-91.7 to -58.3] | -60.6 [-67.7 to -53.3] | -73.9 [-84.6 to -62.5] | -66.7 [-74.2 to -59.4] | -80.0 [-90.5 to -61.5]
  Week 208: number analyzed (Participants) | 37 | 69 | 106 | 131 | 12 | 88 | 14 | 98 | 21
  Week 208 | -87.5 [-97.4 to -82.1] | -81.3 [-88.9 to -72.4] | -83.3 [-89.3 to -78.2] | -92.1 [-96.0 to -88.3] | -75.0 [-86.1 to -56.5] | -85.7 [-90.5 to -80.1] | -74.1 [-85.6 to -55.4] | -84.6 [-88.1 to -78.9] | -81.7 [-90.5 to -66.7]
  Week 260: number analyzed (Participants) | 29 | 56 | 85 | 118 | 9 | 79 | 13 | 85 | 16
  Week 260 | -90.9 [-95.5 to -76.2] | -84.8 [-91.7 to -76.2] | -86.1 [-91.7 to -78.3] | -92.3 [-95.0 to -83.3] | -75.0 [-100.0 to -44.9] | -82.3 [-90.6 to -74.3] | -63.9 [-78.4 to -44.4] | -83.3 [-89.1 to -76.2] | -80.0 [-95.0 to -59.3]

7. Secondary Outcome: Percentage of Participants With Dermatology Life Quality Index (DLQI©) Response (DLQI 0 or 1) Over Time at Weeks 52, 104, 156, 208 and 260
Description: as for outcome 6
Time Frame: Week 52, Week 104, Week 156, Week 208, Week 260
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | AIN150FI | AIN150 FI_AIN300 FI | AIN150FI (NSW+SW) | AIN300 FI | AIN150 SoR | AIN150 SOR_AIN300 FI | AIN300 SoR | AIN300 SoR _ AIN300 FI | AIN300 OL
Number analyzed (Participants) | 77 | 75 | 152 | 168 | 55 | 95 | 60 | 112 | 33
Percentage of participants
  Week 52: number analyzed (Participants) | 77 | 75 | 152 | 165 | 55 | 95 | 60 | 111 | 33
  Week 52 | 59.7 | 57.3 | 58.6 | 72.7 | 32.7 | 34.7 | 28.3 | 41.4 | 54.5
  Week 104: number analyzed (Participants) | 66 | 72 | 138 | 153 | 34 | 91 | 40 | 106 | 30
  Week 104 | 54.5 | 47.2 | 50.7 | 64.7 | 41.2 | 33.0 | 32.5 | 41.5 | 36.7
  Week 156: number analyzed (Participants) | 39 | 75 | 114 | 138 | 16 | 93 | 21 | 109 | 22
  Week 156 | 66.7 | 37.3 | 47.4 | 67.4 | 43.8 | 35.5 | 38.1 | 38.5 | 50.0
  Week 208: number analyzed (Participants) | 37 | 70 | 107 | 132 | 13 | 88 | 14 | 100 | 21
  Week 208 | 62.2 | 52.9 | 56.1 | 70.5 | 30.8 | 62.5 | 42.9 | 59.0 | 52.4
  Week 260: number analyzed (Participants) | 29 | 57 | 86 | 119 | 10 | 79 | 13 | 87 | 16
  Week 260 | 55.2 | 54.4 | 54.7 | 65.5 | 60.0 | 55.7 | 15.6 | 56.3 | 50.0

8. Secondary Outcome: EuroQOL 5-Dimension Health Status Questionnaire (EQ-5D©) Score and Percent Change From Baseline at Weeks 52, 104 and 156
Description: ED-5Q: Participant rated questionnaire to assess health related quality of life in terms of a single utility score. Five domains are assessed mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each with three possible score: 1 indicates no problems, better state of health; 3 indicates worst state of health (example "confined to bed") A visual analog scale (VAS) assesses the health status from 0 (worst possible health state) to 100 (best possible health state)
Time Frame: Baseline, Week 52, Week 104, Week 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | AIN150FI | AIN150 FI_AIN300 FI | AIN150FI (NSW+SW) | AIN300 FI | AIN150 SoR | AIN150 SOR_AIN300 FI | AIN300 SoR | AIN300 SoR _ AIN300 FI | AIN300 OL
Number analyzed (Participants) | 77 | 75 | 152 | 168 | 55 | 95 | 60 | 112 | 33
Percent change
  Week 52: number analyzed (Participants) | 76 | 75 | 151 | 165 | 54 | 93 | 58 | 110 | 33
  Week 52 | 68.8 (137.47) | 57.0 (137.79) | 63.0 (137.30) | 115.8 (666.41) | 40.2 (94.91) | 76.9 (222.97) | 41.3 (140.42) | 98.8 (359.93) | 60.9 (74.18)
  Week 104: number analyzed (Participants) | 65 | 72 | 137 | 153 | 33 | 89 | 40 | 106 | 30
  Week 104 | 58.6 (122.96) | 62.4 (156.21) | 60.6 (140.91) | 118.5 (689.52) | 29.5 (70.63) | 152.9 (902.21) | 46.7 (142.85) | 77.2 (150.86) | 54.3 (84.82)
  Week 156: number analyzed (Participants) | 39 | 75 | 114 | 138 | 14 | 91 | 21 | 107 | 22
  Week 156 | 61.0 (114.81) | 52.1 (115.04) | 55.2 (114.53) | 125.3 (677.23) | 45.1 (102.64) | 140.3 (778.86) | 13.7 (25.16) | 109.5 (373.51) | 68.1 (96.22)

9. Secondary Outcome: Number of Participants With Treatment Emergent Anti-drug Antibodies (ADA)
Description: The development of anti-secunimubab anti-bodies will decrease a participant's ability to respond to secukinumab treatment.
Time Frame: Week 268
Population: The full analysis set (FAS), which consisted of all participants with an observed value, was considered. Only descriptive analysis done.
Measure: Number; unit: Participants
Arm/Group | AIN150FI | AIN150 FI_AIN300 FI | AIN300 FI | AIN150 SoR | AIN150 SOR_AIN300 FI | AIN300 SoR | AIN300 SoR _ AIN300 FI | AIN300 OL
Number analyzed (Participants) | 77 | 75 | 168 | 55 | 95 | 60 | 112 | 33
Participants | 2 | 1 | 3 | 0 | 4 | 0 | 4 | 2

10. Secondary Outcome: Percentage of Patients With Experiencing a Relapse
Description: Relapse is defined as greater than 50% loss of the maximal PASI improvement from baseline.
  PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). A negative mean percentage change indicates improvement.
Time Frame: Week 260
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN150FI | AIN150 FI_AIN300 FI | AIN300 FI | AIN150 SoR | AIN150 SOR_AIN300 FI | AIN300 SoR | AIN300 SoR _ AIN300 FI | AIN300 OL
Number analyzed (Participants) | 77 | 75 | 168 | 55 | 95 | 60 | 112 | 33
Percentage of Participants | 31.2 | 40.0 | 19.6 | 61.8 | 52.6 | 43.3 | 56.3 | 36.4

11. Secondary Outcome: Percentage of Patients With Experiencing a Rebound
Description: Rebound of disease is defined as a worsening of PASI of > 125% of the value at baseline (core study), or new pustular, erythrodermic or more inflammatory psoriasis occurring within 8 weeks of stopping therapy (i.e., if this definition was fulfilled at more than 8 weeks after last study treatment administration, this was defined as rebound like event).
  PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). A negative mean percentage change indicates improvement.
Time Frame: Up to Week 264 (8 weeks post last dose)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AIN150FI | AIN150 FI_AIN300 FI | AIN300 FI | AIN150 SoR | AIN150 SOR_AIN300 FI | AIN300 SoR | AIN300 SoR _ AIN300 FI | AIN300 OL
Number analyzed (Participants) | 77 | 75 | 168 | 55 | 95 | 60 | 112 | 33
Percentage of participants | 11.5 [5.1 to 22.8] | 5.8 [1.9 to 14.9] | 5.0 [2.2 to 10.3] | 9.4 [2.5 to 26.2] | 1.1 [0.1 to 7.0] | 6.9 [1.2 to 24.2] | 10.6 [5.7 to 18.5] | 13.0 [3.4 to 34.7]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 4 years and 7 months.
Description: Consistent with EudraCT disclosure specifications, Novartis has reported under the Serious adverse events fields "number of deaths resulting from adverse events" all those deaths, resulting from serious adverse events that are deemed to be causally related to treatment by the investigator.
Groups:
- Any AIN457 150 mg: Any AIN457 150 mg
- Any AIN457 300 mg: Any AIN457 300 mg
- Any AIN457 Dose: Any AIN457 dose
Arm/Group | Any AIN457 150 mg | Any AIN457 300 mg | Any AIN457 Dose
All-Cause Mortality (participants affected / at risk) | 0/132 | 4/543 | 4/675
Serious Adverse Events (participants affected / at risk) | 25/132 | 119/543 | 144/675
Other Adverse Events (participants affected / at risk) | 93/132 | 449/543 | 542/675
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=132) | Any AIN457 300 mg (N=543) | Any AIN457 Dose (N=675)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 1
LYMPHOID TISSUE HYPERPLASIA (Blood and lymphatic system disorders) | 0 | 1 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 3 | 3
ANGINA UNSTABLE (Cardiac disorders) | 0 | 2 | 2
AORTIC VALVE DISEASE (Cardiac disorders) | 0 | 1 | 1
ARRHYTHMIA (Cardiac disorders) | 0 | 1 | 1
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 1 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 4 | 5
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 1 | 1
BRADYCARDIA (Cardiac disorders) | 0 | 1 | 1
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 | 1 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 1 | 1
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 0 | 2 | 2
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 | 1 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 2 | 2
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 | 1 | 1
CORONARY OSTIAL STENOSIS (Cardiac disorders) | 0 | 1 | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1 | 1
LONG QT SYNDROME (Cardiac disorders) | 0 | 1 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 2 | 2
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1 | 1
MYOCARDITIS (Cardiac disorders) | 0 | 1 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 1 | 1
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 0 | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 1
ANAL INCONTINENCE (Gastrointestinal disorders) | 0 | 1 | 1
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 1 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 1
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 | 1 | 1
LEUKOPLAKIA ORAL (Gastrointestinal disorders) | 1 | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 2 | 2
TOOTHACHE (Gastrointestinal disorders) | 1 | 0 | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 3 | 3
PERIPHERAL SWELLING (General disorders) | 0 | 1 | 1
PYREXIA (General disorders) | 0 | 1 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 3 | 0 | 3
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 2 | 2
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 | 1 | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 | 1 | 1
HEPATITIS ALCOHOLIC (Hepatobiliary disorders) | 0 | 1 | 1
ACUTE HEPATITIS B (Infections and infestations) | 1 | 0 | 1
ACUTE SINUSITIS (Infections and infestations) | 1 | 0 | 1
ANAL ABSCESS (Infections and infestations) | 1 | 0 | 1
APPENDICITIS (Infections and infestations) | 0 | 2 | 2
BURSITIS INFECTIVE STAPHYLOCOCCAL (Infections and infestations) | 0 | 1 | 1
CELLULITIS (Infections and infestations) | 0 | 2 | 2
CHRONIC TONSILLITIS (Infections and infestations) | 0 | 1 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 1 | 1
CYSTITIS (Infections and infestations) | 0 | 1 | 1
EPIDIDYMITIS (Infections and infestations) | 1 | 0 | 1
ERYSIPELAS (Infections and infestations) | 0 | 3 | 3
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 1 | 1
HERPES ZOSTER (Infections and infestations) | 0 | 1 | 1
MENINGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 1 | 1
ORCHITIS (Infections and infestations) | 0 | 1 | 1
OSTEOMYELITIS BACTERIAL (Infections and infestations) | 0 | 1 | 1
PERITONSILLITIS (Infections and infestations) | 0 | 1 | 1
PNEUMONIA (Infections and infestations) | 0 | 6 | 6
SEPSIS (Infections and infestations) | 0 | 1 | 1
SINUSITIS (Infections and infestations) | 0 | 1 | 1
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 | 2 | 2
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1
URINARY TRACT INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 | 1 | 1
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 | 1 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 3 | 3
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 1
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 1 | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1 | 1
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 1 | 1 | 2
LIMB CRUSHING INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
MENISCUS INJURY (Injury, poisoning and procedural complications) | 1 | 1 | 2
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 1 | 1
SPLENIC INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 1
SUBARACHNOID HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 2 | 2
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 3 | 3
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 2 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 2 | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 3 | 3
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1 | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 2 | 2
HEPATIC ENZYME INCREASED (Investigations) | 1 | 3 | 4
LIVER FUNCTION TEST INCREASED (Investigations) | 0 | 1 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 2 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 4
BENIGN LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
BENIGN NEOPLASM OF THYROID GLAND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
BLADDER ADENOCARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
DYSPLASTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 1 | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1 | 1
CAUDA EQUINA SYNDROME (Nervous system disorders) | 0 | 1 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 2 | 2
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 0 | 1 | 1
CUBITAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1 | 1
DIZZINESS (Nervous system disorders) | 0 | 1 | 1
HEADACHE (Nervous system disorders) | 0 | 2 | 2
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1 | 0 | 1
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1 | 1
NERVE COMPRESSION (Nervous system disorders) | 0 | 1 | 1
PERONEAL NERVE PALSY (Nervous system disorders) | 0 | 1 | 1
SCIATICA (Nervous system disorders) | 0 | 1 | 1
SYNCOPE (Nervous system disorders) | 0 | 1 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1 | 1
DEVICE MALFUNCTION (Product Issues) | 0 | 1 | 1
ADJUSTMENT DISORDER (Psychiatric disorders) | 1 | 0 | 1
DELIRIUM (Psychiatric disorders) | 0 | 1 | 1
DEPRESSION (Psychiatric disorders) | 1 | 1 | 2
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 2 | 2
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 1 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 1 | 2
RENAL INFARCT (Renal and urinary disorders) | 1 | 0 | 1
RENAL INJURY (Renal and urinary disorders) | 0 | 1 | 1
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 0 | 1 | 1
URETEROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 1 | 1
URINARY RETENTION (Renal and urinary disorders) | 0 | 1 | 1
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 | 0 | 1
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 1 | 0 | 1
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 | 1 | 1
UTERINE POLYP (Reproductive system and breast disorders) | 0 | 1 | 1
VULVA CYST (Reproductive system and breast disorders) | 0 | 1 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
PULMONARY CAVITATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
RESPIRATORY SYMPTOM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
THORACIC HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
ALCOHOL USE (Social circumstances) | 1 | 0 | 1
AORTIC DILATATION (Vascular disorders) | 0 | 1 | 1
HYPERTENSION (Vascular disorders) | 0 | 1 | 1
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 0 | 1 | 1
VARICOSE VEIN (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=132) | Any AIN457 300 mg (N=543) | Any AIN457 Dose (N=675)
TACHYCARDIA (Cardiac disorders) | 3 | 1 | 4
HYPERTHYROIDISM (Endocrine disorders) | 3 | 0 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 11 | 14
DENTAL CARIES (Gastrointestinal disorders) | 1 | 11 | 12
DIARRHOEA (Gastrointestinal disorders) | 8 | 32 | 40
GASTRITIS (Gastrointestinal disorders) | 4 | 13 | 17
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 | 12 | 15
NAUSEA (Gastrointestinal disorders) | 8 | 9 | 17
TOOTHACHE (Gastrointestinal disorders) | 5 | 21 | 26
VOMITING (Gastrointestinal disorders) | 1 | 16 | 17
FATIGUE (General disorders) | 5 | 16 | 21
NON-CARDIAC CHEST PAIN (General disorders) | 4 | 13 | 17
OEDEMA PERIPHERAL (General disorders) | 3 | 17 | 20
PYREXIA (General disorders) | 3 | 14 | 17
HEPATIC STEATOSIS (Hepatobiliary disorders) | 3 | 9 | 12
SEASONAL ALLERGY (Immune system disorders) | 0 | 16 | 16
BRONCHITIS (Infections and infestations) | 7 | 51 | 58
CELLULITIS (Infections and infestations) | 1 | 15 | 16
CONJUNCTIVITIS (Infections and infestations) | 3 | 19 | 22
FOLLICULITIS (Infections and infestations) | 3 | 25 | 28
FURUNCLE (Infections and infestations) | 2 | 11 | 13
GASTROENTERITIS (Infections and infestations) | 6 | 23 | 29
HERPES ZOSTER (Infections and infestations) | 6 | 13 | 19
INFLUENZA (Infections and infestations) | 12 | 42 | 54
NASOPHARYNGITIS (Infections and infestations) | 31 | 185 | 216
ORAL HERPES (Infections and infestations) | 1 | 19 | 20
PHARYNGITIS (Infections and infestations) | 5 | 28 | 33
RHINITIS (Infections and infestations) | 4 | 22 | 26
SINUSITIS (Infections and infestations) | 8 | 30 | 38
TINEA PEDIS (Infections and infestations) | 3 | 12 | 15
TONSILLITIS (Infections and infestations) | 5 | 20 | 25
TOOTH ABSCESS (Infections and infestations) | 2 | 15 | 17
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 13 | 62 | 75
URINARY TRACT INFECTION (Infections and infestations) | 4 | 23 | 27
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 26 | 26
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1 | 13 | 14
CONTUSION (Injury, poisoning and procedural complications) | 2 | 22 | 24
FALL (Injury, poisoning and procedural complications) | 0 | 11 | 11
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 12 | 13
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 | 19 | 20
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 7 | 10
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 | 15 | 17
HEPATIC ENZYME INCREASED (Investigations) | 5 | 10 | 15
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 20 | 21
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 3 | 12 | 15
GOUT (Metabolism and nutrition disorders) | 0 | 11 | 11
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1 | 12 | 13
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 12 | 12
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 9 | 63 | 72
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9 | 53 | 62
BURSITIS (Musculoskeletal and connective tissue disorders) | 2 | 11 | 13
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 16 | 18
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 15 | 15
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 | 17 | 21
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 | 22 | 30
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 3 | 20 | 23
DIZZINESS (Nervous system disorders) | 3 | 12 | 15
HEADACHE (Nervous system disorders) | 11 | 50 | 61
DEPRESSION (Psychiatric disorders) | 4 | 13 | 17
INSOMNIA (Psychiatric disorders) | 3 | 14 | 17
HAEMATURIA (Renal and urinary disorders) | 5 | 11 | 16
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 51 | 55
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 9
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 31 | 35
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 11 | 11
ACNE (Skin and subcutaneous tissue disorders) | 3 | 3 | 6
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 3 | 6 | 9
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 | 32 | 33
ECZEMA (Skin and subcutaneous tissue disorders) | 6 | 25 | 31
PRURITUS (Skin and subcutaneous tissue disorders) | 9 | 27 | 36
PSORIASIS (Skin and subcutaneous tissue disorders) | 7 | 49 | 56
HYPERTENSION (Vascular disorders) | 8 | 63 | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-04-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT01640951/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT01640951/SAP_001.pdf